CLINICAL TRIAL: NCT06358677
Title: A Phase II, Randomized, Double-Blind, Split-Face of Topical Tretinoin Prophylaxis for Anti-EGFR Induced Skin Toxicity in Patients With Solid Tumors
Brief Title: Topical Tretinoin Prophylaxis for Anti-EGFR Induced Skin Toxicity in Patients With Solid Tumors
Acronym: FACE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCI171997
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Solid Tumor; Locally Advanced Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Tretinoin

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, split-face, phase II study of topical tretinoin prophylaxis for anti-EGFR treatment-induced skin toxicity in patients with locally advanced or metastatic solid tumors.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will apply topical tretinoin to one half of the face and topical moisturizer (placebo) to the other half of the face daily starting the day that anti-EGFR treatment is initiated. The sides of the face tretinoin and moisturizer are applied to will be randomized. Standardized photographs of the face will be obtained at screening and every two weeks from Week 1 Day 1 until after six weeks of treatment. Photographs will be graded by a dermatologist who will be blinded to treatment sidedness. Facial rash severity will be graded using a modified Investigators Global Assessment (IGA) score.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tretinoin half of face (left) and Placebo/Moisturizer other half of the face (right) (Experimental): Randomized, double-blind, split-face. Randomization will determine which side of the face Tretinoin will be applied to (left or right). The other side of the face (left or right) will have placebo applied. All participants will receive both treatment and placebo.
  Interventions: Drug: Topical Tretinoin
- Tretinoin half of face (right) and Placebo/Moisturizer other half of the face (left) (Experimental): Randomized, double-blind, split-face. Randomization will determine which side of the face Tretinoin will be applied to (left or right). The other side of the face (left or right) will have placebo applied. All participants will receive both treatment and placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Topical Tretinoin — Topical tretinoin will be applied to one half of the face, either left or right side. The side the topical tretinoin will be applied to will be randomized.
  Arms: Tretinoin half of face (left) and Placebo/Moisturizer other half of the face (right)
Other: Placebo — A placebo (topical moisturizer) will be applied to the other half of the face, either left or right side. The side the topical tretinoin will be applied to will be randomized.
  Other Names: Topical Moisturizer
  Arms: Tretinoin half of face (right) and Placebo/Moisturizer other half of the face (left)

SUMMARY:
The goal of this clinical trial is to learn if using topical tretinoin will help patients with solid tumors who are experiencing an acneiform rash as a side effect of their treatment.

Researchers will compare the use of tretinoin on one side of the face to the use of a placebo on the other side of the face to see if there is an impact.

DETAILED DESCRIPTION:
The anti-epidermal growth factor receptor (anti-EGFR) agents cetuximab and panitumumab have been shown in numerous trials to be active in patients with metastatic colorectal cancer (mCRC). Current American Society of Clinical Oncology guidelines strongly recommend offering an antiEGFR therapy in combination with chemotherapy to patients with treatment-naïve, left-sided, RAS wild-type mCRC. In addition to colorectal cancer, anti-EGFR agents are also approved for use in the management of head and neck, cutaneous squamous cell, and penile cancers. Novel prophylactic approaches are needed so that more patients can benefit from the survival advantage provided by these drugs without a sacrificing quality of life.

Tretinoin is a vitamin A derivative (all-trans retinoic acid) that has been used by dermatology for more than five decades and is currently approved for the management of moderate to severe acne vulgaris. Initially, tretinoin was recognized as a potential treatment for acne vulgaris based on its comedolytic properties. However, over the past decade tretinoin has been increasingly recognized for its immunomodulatory properties raising the potential for use in dermatologic disorders other than acne vulgaris.

Although the pathogenesis of anti-EGFR associated skin toxicity is still not entirely understood, the clinical presentation shares many similarities with acne vulgaris, and inflammation is felt to play a major role. For this reason, there is interest in the use of tretinoin in the management of anti-EGFR associated rash. Topical tretinoin is associated with minimal transdermal absorption thus making it a viable option for investigation into its use as a prophylactic agent for anti-EGFR associated rash.

This split-face study will utilize a topical moisturizer as a placebo applied to the opposite half of the face as the topical tretinoin. Eucerin, a topical emollient will be used as the placebo in this study. Eucerin is not associated with any significant adverse reactions.

This is a randomized, double-blind, split-face, phase II study of topical tretinoin prophylaxis for anti-EGFR treatment-induced skin toxicity in patients with locally advanced or metastatic solid tumors. Patients will apply topical tretinoin to one half of the face and topical moisturizer (placebo) to the other half of the face daily, starting the day that anti-EGFR treatment is initiated. The sides of the face tretinoin and moisturizer are applied to will be randomized. Standardized photographs of the face will be obtained at screening and every two weeks from Week 1 Day 1 until after six weeks of treatment. Photographs will be graded by a dermatologist who will be blinded to treatment sidedness. Facial rash severity will be graded using a modified Investigators Global Assessment (IGA) score.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged ≥ 18 years
* Histologically confirmed solid tumor.
* Radiologically confirmed locally advanced or metastatic disease.
* Eligible for and willing to receive treatment with panitumumab or cetuximab as standard-of-care.
* ECOG Performance Status ≤ 2.
* Adequate organ function as defined as:

  --Hepatic:
  * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN ----Participants with liver metastases will be allowed to enroll with AST and ALT levels ≤ 5 x ULN.
* Negative pregnancy test for participants who have not undergone surgical sterilization or shown evidence of post-menopausal status. The following age-specific requirements apply:

  --< 50 years of age:
  * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
  * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
  * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

    --≥ 50 years of age:
  * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
  * Had radiation-induced menopause with last menses >1 year ago; or
  * Had chemotherapy-induced menopause with last menses >1 year ago; or
  * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Participants of childbearing potential and participants with a sexual partner of childbearing potential must agree to use a highly effective method of contraception as described in Section 5.4.2.
* Must have recovered from adverse effects of any prior oncologic treatment (e.g. prior surgery, radiotherapy, or other antineoplastic therapy). CTCAE adverse events less than or equal to grade 1 are acceptable. CTCAE adverse events grade 2 or greater may be acceptable as determined by an investigator with appropriate documentation.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Treatment with an anti-EGFR agent within 90 days of registration.
* Pre-existing facial rash that per the treating investigator would preclude the ability to assess response to topical tretinoin.
* The diagnosis of another malignancy within ≤ 2 years before study enrollment, except for those considered to be adequately treated with no evidence of disease or symptoms and/or will not require therapy during the study duration (i.e., basal cell or squamous cell skin cancer, carcinoma in situ of the breast, bladder or of the cervix, or low-grade prostate cancer with Gleason Score ≤ 6).
* Any other condition that would, in the Investigator's judgment, contraindicate the participant's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Systemic active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C.

  --Note: Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Participants positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Medical, psychiatric, cognitive, or other conditions that may compromise the participant's ability to understand the participant information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity to investigational product or any component in its formulations (CTCAE v5.0 Grade ≥ 3).
* Participants taking prohibited medications as described in Section 6.8.2. A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
The maximum difference in modified Investigators Global Assessment (IGA) score between the treated and untreated sides of the face at any assessment. | up to 6 weeks from the initiation of study therapy
  Effect of topical tretinoin on anti-EGFR induced acneiform rash. Rash will be scored from 0-4 with 0 being clear skin and 4 being a severe rash.

SECONDARY OUTCOMES:
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE version 5.0 and the modified IGA), seriousness, duration, and relationship to study treatment. | up to 6 weeks from the initiation of study therapy
  Proportion of acneiform rash per CTCAE v5.0
Proportion of acneiform rash per CTCAE v5.0 | up to 6 weeks from the initiation of study therapy
  To assess the safety and tolerability of topical tretinoin in the study population.
  This outcome measure will report the frequency of acneiform rash as defined by the NIH CTCAE, version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nevala-Plagemann, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Cutsem E, Kohne CH, Lang I, Folprecht G, Nowacki MP, Cascinu S, Shchepotin I, Maurel J, Cunningham D, Tejpar S, Schlichting M, Zubel A, Celik I, Rougier P, Ciardiello F. Cetuximab plus irinotecan, fluorouracil, and leucovorin as first-line treatment for metastatic colorectal cancer: updated analysis of overall survival according to tumor KRAS and BRAF mutation status. J Clin Oncol. 2011 May 20;29(15):2011-9. doi: 10.1200/JCO.2010.33.5091. Epub 2011 Apr 18. PMID 21502544
- [Background] Berlin J, Posey J, Tchekmedyian S, Hu E, Chan D, Malik I, Yang L, Amado RG, Hecht JR. Panitumumab with irinotecan/leucovorin/5-fluorouracil for first-line treatment of metastatic colorectal cancer. Clin Colorectal Cancer. 2007 Mar;6(6):427-32. doi: 10.3816/CCC.2007.n.011. PMID 17531105
- [Background] Kohne CH, Hofheinz R, Mineur L, Letocha H, Greil R, Thaler J, Fernebro E, Gamelin E, Decosta L, Karthaus M. First-line panitumumab plus irinotecan/5-fluorouracil/leucovorin treatment in patients with metastatic colorectal cancer. J Cancer Res Clin Oncol. 2012 Jan;138(1):65-72. doi: 10.1007/s00432-011-1061-6. Epub 2011 Sep 30. PMID 21960318
- [Background] Watanabe J, Muro K, Shitara K, Yamazaki K, Shiozawa M, Ohori H, Takashima A, Yokota M, Makiyama A, Akazawa N, Ojima H, Yuasa Y, Miwa K, Yasui H, Oki E, Sato T, Naitoh T, Komatsu Y, Kato T, Hihara M, Soeda J, Misumi T, Yamamoto K, Akagi K, Ochiai A, Uetake H, Tsuchihara K, Yoshino T. Panitumumab vs Bevacizumab Added to Standard First-line Chemotherapy and Overall Survival Among Patients With RAS Wild-type, Left-Sided Metastatic Colorectal Cancer: A Randomized Clinical Trial. JAMA. 2023 Apr 18;329(15):1271-1282. doi: 10.1001/jama.2023.4428. PMID 37071094
- [Background] Nevala-Plagemann C, Iyengar S, Trunk AD, Pappas L, Haaland B, Garrido-Laguna I. Treatment Trends and Clinical Outcomes of Left-Sided RAS/RAF Wild-Type Metastatic Colorectal Cancer in the United States. J Natl Compr Canc Netw. 2022 Feb 4;20(3):268-275. doi: 10.6004/jnccn.2021.7079. PMID 35120306
- [Background] Ciliberto D, Staropoli N, Caglioti F, Chiellino S, Ierardi A, Ingargiola R, Botta C, Arbitrio M, Correale P, Tassone P, Tagliaferri P. The best strategy for RAS wild-type metastatic colorectal cancer patients in first-line treatment: A classic and Bayesian meta-analysis. Crit Rev Oncol Hematol. 2018 May;125:69-77. doi: 10.1016/j.critrevonc.2018.03.003. Epub 2018 Mar 9. PMID 29650279
- [Background] Morris VK, Kennedy EB, Baxter NN, Benson AB 3rd, Cercek A, Cho M, Ciombor KK, Cremolini C, Davis A, Deming DA, Fakih MG, Gholami S, Hong TS, Jaiyesimi I, Klute K, Lieu C, Sanoff H, Strickler JH, White S, Willis JA, Eng C. Treatment of Metastatic Colorectal Cancer: ASCO Guideline. J Clin Oncol. 2023 Jan 20;41(3):678-700. doi: 10.1200/JCO.22.01690. Epub 2022 Oct 17. PMID 36252154
- [Background] Lacouture ME, Anadkat M, Jatoi A, Garawin T, Bohac C, Mitchell E. Dermatologic Toxicity Occurring During Anti-EGFR Monoclonal Inhibitor Therapy in Patients With Metastatic Colorectal Cancer: A Systematic Review. Clin Colorectal Cancer. 2018 Jun;17(2):85-96. doi: 10.1016/j.clcc.2017.12.004. Epub 2017 Dec 13. PMID 29576427
- [Background] Lacouture ME, Mitchell EP, Piperdi B, Pillai MV, Shearer H, Iannotti N, Xu F, Yassine M. Skin toxicity evaluation protocol with panitumumab (STEPP), a phase II, open-label, randomized trial evaluating the impact of a pre-Emptive Skin treatment regimen on skin toxicities and quality of life in patients with metastatic colorectal cancer. J Clin Oncol. 2010 Mar 10;28(8):1351-7. doi: 10.1200/JCO.2008.21.7828. Epub 2010 Feb 8. PMID 20142600
- [Background] Zaenglein AL, Pathy AL, Schlosser BJ, Alikhan A, Baldwin HE, Berson DS, Bowe WP, Graber EM, Harper JC, Kang S, Keri JE, Leyden JJ, Reynolds RV, Silverberg NB, Stein Gold LF, Tollefson MM, Weiss JS, Dolan NC, Sagan AA, Stern M, Boyer KM, Bhushan R. Guidelines of care for the management of acne vulgaris. J Am Acad Dermatol. 2016 May;74(5):945-73.e33. doi: 10.1016/j.jaad.2015.12.037. Epub 2016 Feb 17. PMID 26897386
- [Background] Baldwin HE, Nighland M, Kendall C, Mays DA, Grossman R, Newburger J. 40 years of topical tretinoin use in review. J Drugs Dermatol. 2013 Jun 1;12(6):638-42. PMID 23839179
- [Background] Schmidt N, Gans EH. Tretinoin: A Review of Its Anti-inflammatory Properties in the Treatment of Acne. J Clin Aesthet Dermatol. 2011 Nov;4(11):22-9. PMID 22125655
- [Background] Holcmann M, Sibilia M. Mechanisms underlying skin disorders induced by EGFR inhibitors. Mol Cell Oncol. 2015 Jun 1;2(4):e1004969. doi: 10.1080/23723556.2015.1004969. eCollection 2015 Oct-Dec. PMID 27308503
- [Background] Vezzoli P, Marzano AV, Onida F, Alessi E, Galassi B, Tomirotti M, Berti E. Cetuximab-induced acneiform eruption and the response to isotretinoin. Acta Derm Venereol. 2008;88(1):84-6. doi: 10.2340/00015555-0330. No abstract available. PMID 18176767
- [Background] Gutzmer R, Werfel T, Mao R, Kapp A, Elsner J. Successful treatment with oral isotretinoin of acneiform skin lesions associated with cetuximab therapy. Br J Dermatol. 2005 Oct;153(4):849-51. doi: 10.1111/j.1365-2133.2005.06835.x. No abstract available. PMID 16181478
- [Background] Kizilyel O, Metin MS, Elmas OF, Cayir Y, Aktas A. Effects of oral isotretinoin on lipids and liver enzymes in acne patients. Cutis. 2014 Nov;94(5):234-8. PMID 25474452
- [Background] van Hoogdalem EJ. Transdermal absorption of topical anti-acne agents in man; review of clinical pharmacokinetic data. J Eur Acad Dermatol Venereol. 1998 Sep;11 Suppl 1:S13-9; discussion S28-9. doi: 10.1111/j.1468-3083.1998.tb00902.x. PMID 9891904
- [Background] Kligman AM, Grove GL, Hirose R, Leyden JJ. Topical tretinoin for photoaged skin. J Am Acad Dermatol. 1986 Oct;15(4 Pt 2):836-59. doi: 10.1016/s0190-9622(86)70242-9. PMID 3771853
- [Background] Griffiths CE, Kang S, Ellis CN, Kim KJ, Finkel LJ, Ortiz-Ferrer LC, White GM, Hamilton TA, Voorhees JJ. Two concentrations of topical tretinoin (retinoic acid) cause similar improvement of photoaging but different degrees of irritation. A double-blind, vehicle-controlled comparison of 0.1% and 0.025% tretinoin creams. Arch Dermatol. 1995 Sep;131(9):1037-44. PMID 7544967
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009